CLINICAL TRIAL: NCT06151691
Title: Explorations of Cell-free DNA Multi-omics Technology in Detection of Minimal Residual Disease and Disease Prognosis After Surgery in Early Pancreatic Ductal Adenocarcinoma: A Single-center, Prospective, Observational Case Study
Brief Title: Assessment of Early Pancreatic Cancer Prognosis by Minimal Residual Disease Using Multi-omics Approach
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Collaborators: Shanghai Weihe Medical Laboratory Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xian-Jun Yu, M.D., Ph.D., Fudan University
Other Study IDs: PC-MRD
Record Dates: First submitted 2023-11-22; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cfDNA and tumor tissue DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case-Cancer arm: Blood collection and Pancreatic ductal adenocarcinoma minimal residual disease detection test
  Interventions: Other: Blood collection and Pancreatic ductal adenocarcinoma minimal residual disease detection test

INTERVENTIONS:
Other: Blood collection and Pancreatic ductal adenocarcinoma minimal residual disease detection test — Blood samples of participants meet the inclusion/exclusion criteria will be collected.
  Pancreatic ductal adenocarcinoma minimal residual disease detection test.

SUMMARY:
This trial aims to develop a minimal residual disease (MRD) detection model for predicting recurrence of patients with stage I-II pancreatic ductal adenocarcinoma after surgery and adjuvant therapy, based on cfDNA fragmentation and methylation signal.

DETAILED DESCRIPTION:
The entire study is divided into two stages. Stage one is the enrollment period. 51 subjects with pancreatic ductal adenocarcinoma in stages I-II who have not received neoadjuvant therapy and have undergone radical surgery were enrolled. Blood samples at the time point before surgical treatment (T0) were collected and fresh tissue specimens (cancerous tissue and adjacent normal tissue) were collected. Blood samples were subjected to methylation, fragment group, and CNV multi-omics testing, and tissue samples were subjected to target methylation area testing. Stage two is the follow-up period. Blood samples from the fifth week after surgery to before adjuvant therapy (T1) and blood samples from 4-8 weeks after adjuvant therapy (T2) were collected. Blood samples were subjected to methylation, fragment group, and CNV multi-omics testing with different techniques. The subjects were followed up for 1.5 years. According to progression and recurrence, the subjects were divided into progression group and non-progression group. Methylation and multi-omics prognosis models were trained and compared for their performance in residual detection and recurrence prediction.

ELIGIBILITY:
Inclusion criteria:

1. Patients with clinically and/or pathologically diagnosis of stage I/II pancreatic ductal adenocarcinoma;
2. Aged ≥ 40 years and < 75 years, both sexes;
3. Patients receive radical resection with curative intent, followed by adjuvant therapy;
4. Tumour size not less than 1 cm * 1 cm * 1 cm and be able to provide surgical tissue samples for molecular testing after pathological evaluation;
5. Eastern Cooperative Oncology Group (ECOG) score of 0-2;
6. Negative margins (R0 or R1) by naked eye or no recurrence/metastasis detected on imaging after surgery or before adjuvant therapy, and CA 19-9<37 U/ml;
7. Patients understand and voluntarily sign the informed consent form and follow the sampling, assessment and visit requirements of this study.

Exclusion criteria:

1. Pregnant and lactating (by self-report);
2. Any tumor history of malignancies;
3. Positive cutting margins (R2);
4. Received neoadjuvant therapy before surgery;
5. Not be able to receive radical surgery;
6. Organ transplantation history;
7. Organ dysfunction (moderate or severe renal impairment with absolute centrocyte count < 1.0 x 10^9/L, platelet count < 75 x 10^9/L, haemoglobin < 80 g/L, AST/ALT > 2.5 times upper limit of normal);
8. Other conditions deemed unsuitable for enrollment by the investigator.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be recruited from clinic and medical centers. Participants are defined as new diagnosis cancer patients with pancreatic ductal adenocarcinoma. Demographic and cancer risk-related characteristics (eg, age, gender, smoking status, diabetes) will be collected from all enrolled subjects.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
1.5-year disease-free survival | 18 months
  1.5-year disease-free survival of patients with pancreatic ductal adenocarcinoma receiving post-operative adjuvant chemotherapy.

SECONDARY OUTCOMES:
Sensitivity of the multi-omics prognostic model | 18 months
  Sensitivity of the multi-omics prognostic model for pancreatic ductal adenocarcinoma based on cfDNA methylation, fragmentation group, and CNV features in patients with recurrence at 95% confidence interval
Specificity of the multi-omics prognostic model | 18 months
  Specificity of the multi-omics prognostic model for pancreatic ductal adenocarcinoma patients without recurrence at 95% confidence intervals.
Area under the receiver operating characteristic curve (AUROC) of the multi-omics prognostic model | 18 months
  Area under the receiver operating characteristic curve (AUROC) of the multi-omics prognostic model for predicting patient recurrence of pancreatic ductal adenocarcinoma at 95% confidence intervals.
Sensitivity of the multi-omics prognostic model in different subgroups | 18 months
  Sensitivity of the multi-omics prognostic model for predicting pancreatic ductal adenocarcinoma recurrence in different subgroups (age, underlying medical history, tumour differentiation, tumour diameter, etc.) at 95% confidence intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pancreatic and Hepatobiliary Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University; 270 Dong An Road, Shanghai 200032, China, Shanghai, China

IPD SHARING:
Plan to Share IPD: No